CLINICAL TRIAL: NCT04139759
Title: Randomized Controlled Quasi-experimental
Brief Title: THE EFFECT OF HAND AND FOOT MASSAGE ON FATIGUE IN HEMODIALYSIS PATIENTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Sultan ÇEÇEN, lecturer, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: massage
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Hemodialysis Patients
Keywords: Nursing; Hemodialysis; Fatigue; Hand massage; Foot massage
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hand massage group (Experimental): In the hand massage group (n = 28), hand massage was applied to the hand without fistula for 8 minutes, 3 times a week, for 4 weeks.
  Interventions: Other: hand massage
- Foot massages group (Experimental): Foot massages were applied to both feet of the patients in the foot massage group (n = 28), 3 times a week, for 4 weeks and patting and kneading movements were repeated 3-4 times.
  Interventions: Other: foot massage
- control group (No Intervention): The patients in the control group (n = 28) were not administered except nursing interventions in the HD unit.

INTERVENTIONS:
Other: hand massage — In the hand massage group (n = 28), hand massage was applied to the hand without fistula for 8 minutes, 3 times a week, for 4 weeks.
  Arms: hand massage group
Other: foot massage — Foot massages were applied to both feet of the patients in the foot massage group (n = 28), 3 times a week, for 4 weeks and patting and kneading movements were repeated 3-4 times.
  Arms: Foot massages group

SUMMARY:
Hemodialysis patients face many problems related to disease and treatment, fatigue is stated as the most common of these problems. Therefore, The aim of this study is to examine the effect of hand massage and foot massage on fatigue in hemodialysis patients.

DETAILED DESCRIPTION:
In parallel with the recent technological advances in medicine, increasing the possibilities of diagnosis and treatment of diseases has increased the average life expectancy and the incidence of chronic diseases. Chronic renal failure (CRF), which is one of the increasing chronic diseases, has become an important public health problem due to its negative impact on quality of life both in the world and in our country, high morbidity, mortality and treatment costs. According to the Joint Report of the Turkish Ministry of Health and Turkish Nephrology Association; by the end of 2016, Renal Replacement Therapy (RRT) applied total 74,475 patients (including pediatric patients), RRT is applied and while the most common form of treatment has been found to be hemodialysis treatment with 76.12%. Unless a successful renal transplantation is performed, hemodialysis treatment required to be performed until the end of life and provides a longer life, but it also causes biological, psychological, social and economical problems arising from treatment. Fatigue, which often related to problems with its biological dimension, reduces the quality of life by adversely negatively affecting individual's daily life activities.

ELIGIBILITY:
Inclusion Criteria:

* - Taking HD therapy, in the dialysis unit of a public hospital in Turkey, between October 19, 2018 - February 11, 2019,
* Agree to participate in the study with a written permission,
* Over the age of 18,
* Open to communication with complete orientation,
* Speaks and understands Turkish
* Receiving HD treatment 3 times a week for 6 months and longer,
* No loss of sensation, mass, fracture or ingrown toenail (onyxis),
* In the lower extremities; without pathological and tumoral disease, phlesis, embolism and no bleeding disorder related to amputation, fracture, infection, wound, skin disease, muscle and bones,
* Patients with a Standardized Mini Mental Test (SMMT) score of 24 or more, in patients older than 65 years,

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Pre-Hemodialysis / 1st Measurement | first day
  In addition to verbal and written information, the first measurements were obtained by applying the Patient Presentation Form, Visual Similarity Scale for Fatigue to the patients who were taken to hand massage, foot massage and control groups before HD treatment. In 1990, Lee et al. developed the Visual Similarity Scale for Fatigue, consisting of 18 items, to determine fatigue. The items 1, 2, 3, 4, 5, 11, 12, 13, 14, 15, 16, 17, 18 of the scale included fatigue subcomponent and 6, 7, 8, 9,10 items belong to the energy subcomponent. The Visual Similarity Scale for Fatigue consists of 10 cm lines, the most positive expression at one end and the negative expression at the other end of the line. The high score of the fatigue subcomponent, the low score of the energy subcomponent, shows that the severity of fatigue is high.

SECONDARY OUTCOMES:
2 Weeks Later /2nd Measurement | fifteenth day
  At the end of the second week of the hand massage and foot massage applications, the second measurements were obtained by reapplying the Visual Similarity Scale for Fatigue scale to all three groups.In 1990, Lee et al. developed the Visual Similarity Scale for Fatigue, consisting of 18 items, to determine fatigue. The items 1, 2, 3, 4, 5, 11, 12, 13, 14, 15, 16, 17, 18 of the scale included fatigue subcomponent and 6, 7, 8, 9,10 items belong to the energy subcomponent. The Visual Similarity Scale for Fatigue consists of 10 cm lines, the most positive expression at one end and the negative expression at the other end of the line. The high score of the fatigue subcomponent, the low score of the energy subcomponent, shows that the severity of fatigue is high.

OTHER OUTCOMES:
4 Weeks Later/ 3rd Measurement | thirtieth day
  At the end of the third week of the hand massage and foot massage applications, the third measurements were obtained by reapplying the Visual Similarity Scale for Fatigue scale to all three groups.In 1990, Lee et al. developed the Visual Similarity Scale for Fatigue, consisting of 18 items, to determine fatigue. The items 1, 2, 3, 4, 5, 11, 12, 13, 14, 15, 16, 17, 18 of the scale included fatigue subcomponent and 6, 7, 8, 9,10 items belong to the energy subcomponent. The Visual Similarity Scale for Fatigue consists of 10 cm lines, the most positive expression at one end and the negative expression at the other end of the line. The high score of the fatigue subcomponent, the low score of the energy subcomponent, shows that the severity of fatigue is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Batman Regional State Hospital, Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
de-identified individual participate data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Astroth KS, Russell CL, Welch JL. Non-pharmaceutical fatigue interventions in adults receiving hemodialysis: a systematic review. Nephrol Nurs J. 2013 Sep-Oct;40(5):407-27; quiz 428. PMID 24308108
- [Result] Ahmadidarrehsima S, Mohammadpourhodki R, Ebrahimi H, Keramati M, Dianatinasab M. Effect of foot reflexology and slow stroke back massage on the severity of fatigue in patients undergoing hemodialysis: A semi-experimental study. J Complement Integr Med. 2018 Sep 28;15(4). doi: 10.1515/jcim-2017-0183. PMID 30265652